CLINICAL TRIAL: NCT06464081
Title: Tongue Muscular Assessment in Children (TMAC) - Reproducibility Testing
Status: Recruiting | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, William Poncin, Prof., Université Catholique de Louvain
Other Study IDs: TMAC-reprod
Record Dates: First submitted 2024-06-12; First posted 2024-06-18 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Healthy
Keywords: tongue; motor skills
MeSH Terms: interventions — Anthropometry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inter-rater reliability and intra-rater reliability: Tongue protrusion, elevation and swallowing measurements will be assessed at three time points, each interspersed by a one-week to one-month interval.
  Assessments will be conducted by the same rater during two of these time points, whereas another independent rater will conduct the assessments of the third time point.
  Interventions: Other: Sleep quality assessment; Other: Anthropometry; Other: Tongue strength assessment; Other: Tongue endurance assessment; Other: Orofacial praxis assessment

INTERVENTIONS:
Other: Sleep quality assessment — 1. Pediatric Sleep Questionnaire.
Other: Anthropometry — 2. Anthropometric data : 2.1 Height; 2.2 Weight; 2.3 Maximal mouth opening; 2.4 Maximal mouth opening with tongue to palate The measures 2.3 and 2.4 will be realized via the Quick Tongue-Tie assessment tool
Other: Tongue strength assessment — 3. Tongue pressure while swallowing. 4. Tongue peak pressure during tongue elevation. 5. Tongue peak pressure during tongue protrusion. These measures will be realized via the IOPI (Iowa Oral Performance Instrument) device.
Other: Tongue endurance assessment — 6. The tongue endurance during tongue elevation. 7. The tongue endurance during tongue protrusion. These measures will be realized via the IOPI (Iowa Oral Performance Instrument) device and a timer.
Other: Orofacial praxis assessment — 8. Motricité Bucco-Linguo-Faciale (MBLF) test.

SUMMARY:
This study aims to assess intra-rater and inter-rater reliability in measuring tongue motor skills in children.

DETAILED DESCRIPTION:
Several motor skills of the tongue can be described: tongue elevation, swallowing, and protrusion. They are all relevant for a wide array of disorders, including neurological, musculoskeletal, and respiratory conditions. An ongoing study by our team is attempting to collect normative data on these motor skills in a pediatric cohort (NCT06166680). From this ongoing study, 56 subjects will be selected to assess the intra-rater and inter-rater reliability in measuring these motor skills.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 4 and 17 years old

Exclusion Criteria:

* Eating disorder
* Dysphagia
* Cardiorespiratory disorder
* Neurological disorder (including neuromuscular disorders)
* Previous or ongoing obstructive sleep apnea-hypopnea syndrome
* Previous or ongoing cancer of the head or neck
* Previous oral or pharyngeal surgery (except for the surgical removal of wisdom teeth)
* Cranial, oral or upper airway malformation (ex.: nasal cavities, pharynx)
* Previous or ongoing orthodontic treatment (e.g. braces)
* More than 33% of positive answers to the Pediatric Sleep Questionnaire (≥ 8/22)

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children aged between 4 and 17 years old
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Test-retest reproducibility of tongue peak pressure | Measured at baseline, and then at two other time points. These three time points will each be interspersed by a one-week to one-month interval
  Tongue peak pressure during elevation and protrusion movements will be measured. The inter-rater and intra-rater reliability of these measures will be computed.

SECONDARY OUTCOMES:
Test-retest reproducibility of tongue endurance | Measured at baseline, and then at two other time points. These three time points will each be interspersed by a one-week to one-month interval
  Tongue endurance during elevation and protrusion movements will be measured. The inter-rater and intra-rater reliability of these measures will be computed.
Test-retest reproducibility of tongue pressure during swallowing | Measured at baseline, and then at two other time points. These three time points will each be interspersed by a one-week to one-month interval
  Tongue pressure during swallowing will be measured. The inter-rater and intra-rater reliability of these measures will be computed.
Test-retest reproducibility of tongue mobility restriction | Measured at baseline, and then at two other time points. These three time points will each be interspersed by a one-week to one-month interval
  Assessed through the ratio between maximal mouth opening and maximal mouth opening with tongue to palate. The inter-rater and intra-rater reliability of these measures will be computed.
Test-retest reproducibility of orofacial praxis | Measured at baseline, and then at two other time points. These three time points will each be interspersed by a one-week to one-month interval
  Orofacial praxis will be assessed. The inter-rater and intra-rater reliability of this measure will be computed.

CONTACTS AND LOCATIONS:
Overall Officials: William Poncin, Prof, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Woluwe-Saint-Lambert, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No